CLINICAL TRIAL: NCT04286009
Title: Pathogenesis and Mechanisms of Mitral Annular Calcification
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Other Study IDs: 19-011417
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Mitral Annulus Calcification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
  Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are testing blood or mitral valve tissue to better understand the reasons why Mitral Annular Calcification (MAC) develops in patients with heart disease.

DETAILED DESCRIPTION:
The aim is to test the hypothesis that Endothelial Progenitor Cells osteoblastic phenotype (EPC-OCNs) play a significant role in the process of Mitral Annular Calcification (MAC) as prognostic markers of calcific cardiac valves.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of MAC and patients coming to the Valve Clinic without MAC diagnosis Patients who will undergo surgery, either standard surgical MVR or trans-atrial TMVR, with diagnosis of MAC or without diagnosis of MAC

Exclusion Criteria:

* Subjects unwilling to participate or to provide consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects referred to the Mayo Clinic valve clinic, with or without MAC. Also, subjects undergoing surgery, either standard surgical MVR or trans-atrial TMVR.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Prognostic markers of calcific cardiac valves | Baseline
  Measured by Endothelial Progenitor Cells osteoblastic phenotype (EPC-OCNs) in Mitral Annular Calcification (MAC)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No